CLINICAL TRIAL: NCT06506266
Title: A Randomized, Double-blind, Single-site, Two-way Crossover Phase 1 Study to Assess the Effect of Repeated Doses of Test Propellant (HFA-152a) on Mucociliary Clearance as Compared to Reference Propellant (HFA-134a) in Healthy Male and Female Participants
Brief Title: Study of the Effect of HFA-152a and HFA-134a Propellants on Mucociliary Clearance in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 221781
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Asthma
Keywords: HFA-152a; HFA-134a; Crossover; MCC
MeSH Terms: conditions — Asthma | interventions — norflurane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HFA-152a followed by HFA-134a (Experimental)
  Interventions: Other: HFA-152a; Other: HFA-134a; Other: Radiolabeled saline solution
- HFA-134a followed by HFA-152a (Experimental)
  Interventions: Other: HFA-152a; Other: HFA-134a; Other: Radiolabeled saline solution

INTERVENTIONS:
Other: HFA-152a — HFA-152a is administered via oral inhalation
Other: HFA-134a — HFA-134a is administered via oral inhalation
Other: Radiolabeled saline solution — Radiolabeled saline solution is administered via oral inhalation

SUMMARY:
The main goal of the study is to assess the effect of the administration of reference propellant [HFA-134a (1,1,1,2 - Tetrafluoroethane)] and test propellant [HFA-152a (1 - Difluoroethane)] in healthy adults on mucociliary clearance (MCC).

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all following criteria apply:

* Male or Female, age 30 to 55 years
* Body Mass Index (BMI): 18.0 to 32.0 kg/m2, inclusive, at screening
* Weight: ≥50 kg
* Nonsmokers or ex-smokers for more than 6 months with a smoking history of <10 pack years
* Status: healthy participants
* Spirometry data.

  * Forced Expiratory Volume in 1 second (FEV1) ≥80% of predicted values.
  * FEV1: Forced vital capacity (FVC) ratio >70%.
* Females must be of nonchildbearing potential, and agree not to donate eggs (ova, oocytes) for the purpose of reproduction during the study intervention period and at least 30 days after the last dose of study intervention.
* Male participants are eligible to participate if they agree to:

  * Refrain from donating sperm
  * Either be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent
  * Or must agree to use a male condom when having sexual intercourse with a woman of childbearing potential (WOCBP) who is not currently pregnant. The female partner should additionally use a highly effective contraceptive method with a failure rate of <1% per year.
* All prescribed medication must have been stopped at least 30 days prior to admission to the clinical research centre based on investigator judgment. An exception is made for Hormonal Replacement Therapy (HRT), and occasional paracetamol which may be used throughout the study.
* Capable of giving written informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Capable of using inhaler device with no physical or other issues which would impair the participant's ability to successfully use a metered dose inhaler (MDI) inhaler as instructed in this study.
* Ability to comply with the protocol. Participants have capacity and no issues which would impair their ability to comply with all aspects of the protocol during the study

Exclusion Criteria:

Participants who meet any of the following exclusion criteria at screening will not be eligible to participate in the study:

* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 millisievert (mSv) in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker shall participate in the study.
* History or presence of any form of asthma, including childhood asthma and exercise induced asthma.
* Respiratory disorders other than asthma. A history of respiratory diseases to include (but not limited to): pneumothorax, pulmonary fibrotic disease, bronchopulmonary dysplasia, chronic bronchitis, cystic fibrosis, bronchiectasis, interstitial lung disease, emphysema, Chronic obstructive pulmonary disease (COPD), tuberculosis, known alpha 1 antitrypsin deficiency and other respiratory abnormalities other than asthma that, in the opinion of the investigator, could put the participant at risk through study participation or could affect the study analyses and data interpretation.
* Recent history of mild conditions potentially affecting Mucociliary clearance (MCC) (viral infections, cough, cold, active hay fever etc.) in the last 14 days.
* Recent use of drugs for treating conditions potentially affecting MCC (viral infections, cough, cold, etc.) in the last 30 days.
* Vaccine(s) within 2 weeks prior to admission or plans to receive such vaccines during the study.
* Current enrolment or past participation in this clinical study.
* Positive human immunodeficiency virus (HIV) antibody test.
* Regular use of known drugs of abuse, including Tetrahydrocannabinol (THC).
* Average intake of more than 21 units of alcohol per week in males and 14 units per week in females (clinical site standard: unit of alcohol equals approximately 250 mL of beer, 100 mL of wine, or 35 mL of spirits) based on breath alcohol test.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-07-29 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Area under the percent radiolabeled particle retention-time curve up to 4 hours [AUC(0-4h)] following administration of nebulized inhalation of saline solution | Up to 4 hours on Day 7

SECONDARY OUTCOMES:
Percent radiolabeled particle retention at 1 hour after nebulized inhalation of saline solution | 1 hour after inhalation of saline solution on Day 7
Percent radiolabeled particle retention at 1.5 hours after nebulized inhalation of saline solution | 1.5 hours after inhalation of saline solution on Day 7
Percent radiolabeled particle retention at 3 hours after nebulized inhalation of saline solution | 3 hours after inhalation of saline solution on Day 7
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to 56 days

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/